CLINICAL TRIAL: NCT01299051
Title: Steps to Health: Targeting Obesity in the Health Care Workplace
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Duke University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None
Other Study IDs: Pro00010727; R01HD06578 (Other Grant/Funding Number: National Institute of Occupational Safety and Health)
Record Dates: First submitted 2011-02-03; First posted 2011-02-18 (Estimated); Last update posted 2016-03-08 (Estimated); Status verified 2016-03

CONDITIONS: Overweight; Obese
Keywords: Weight Management; Employee Health
MeSH Terms: conditions — Overweight; Obesity

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Steps to Health (Active Comparator): Steps to Health worksite weight management program at Duke.
  Interventions: Behavioral: Steps to Health
- Steps to Health Plus! (Experimental): Steps to Health Plus! worksite weight management program at Duke. Also known as Pathways to Change.
  Interventions: Behavioral: Steps to Health Plus!
- Observational Comparison (No Intervention): Observational comparison group consisting of employees who are eligible for the study but do not take part will also be used in analyses (approximately 1500 subjects).

INTERVENTIONS:
Behavioral: Steps to Health — Steps to Health (STH): The STH curriculum is a 12-month educational program targeting obese employees for healthy lifestyle changes for weight loss. The program includes:
  * Face-to-face visit with counselor during Month 1 to set specific health goals.
  * Telephone counseling at 6 and 12 months, coupled with biometric feedback sessions.
  * Monthly generic health education materials sent via e-mail.
  * Incentives (up to 1,000 STH dollars [$100]) to take part in the program assessments.
  Other Names: STH
  Arms: Steps to Health
Behavioral: Steps to Health Plus! — The STH+ intervention is an intensive 12-month behavioral intervention targeting obese employees. It is stage-based and works with the participant at his/her level of readiness to change using counseling based on motivational interviewing. STH+ includes:
  * Face-to-face visit with counselor at Month 1
  * Meeting with exercise physiologist in Month 2
  * Monthly counseling sessions (in-person in Months 3, 6, 9 and 12, others via telephone)
  * Meeting with exercise physiologist during Month 5
  * Quarterly biometric feedback (Months 3, 6, 9, and 12)
  * Incentives (up to 1,000 STH dollars [$100]) to take part in the program assessments.
  Other Names: STH+, PTC
  Arms: Steps to Health Plus!

SUMMARY:
The proposal of this study is to compare the effectiveness of two worksite weight management programs at Duke: Steps to Health (STH) ('usual standard of care') and the more extensive Steps to Health Plus! (STH+). We have added an additional follow-up, by invitation only, for participants in the study who agreed to be contacted for future research.

DETAILED DESCRIPTION:
Steps to Health and Steps to Health Plus! aim to help Duke employees achieve weight loss and maintain healthy weights. We will be following participants in these programs over a two year period. These two groups will be compared with an observational comparison group of employees who meet eligibility criteria but do not take part in the randomized controlled trial. We will assess whether the two programs decrease obesity-related injuries in the workplace and estimate the net costs of the two programs relative to their effectiveness more broadly.

In the additional follow-up, we will be assessing factors that may be related to program success. This will include a survey as well as some focus group data.

ELIGIBILITY:
Inclusion Criteria:

* Completion of a Health Risk Assessment
* BMI ≥ 30
* Able to read and understand study materials which are presented in English
* No plans to leave Duke in the next year
* Enrolled in one of the Duke health plans
* Not currently pregnant

Exclusion Criteria:

* Enrolled in the other available individual intervention programs (hypertension, cholesterol or pre-diabetes)
* Enrolling in one of the LFL weight management programs in order to qualify for bariatric surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 550 (Actual)
Dates: Start 2011-01; Primary Completion 2014-10 (Actual); Study Completion 2016-03 (Actual)

PRIMARY OUTCOMES:
Weight loss | ~1-2 years post baseline
  Determine whether employees participating in STH+ will lose significantly more body mass than participants in STH.

SECONDARY OUTCOMES:
Improvement in level of physical activity | ~1-2 years post baseline.
  Determine whether employees participating in STH+ will experience greater improvements level or amount of physical activity than employees in STH.
Relative impact of the different programs | ~1-2 years post baseline
  Determine the relative impact of STH+ and STH on 1) reduction in workplace injuries and associated costs, 2) health care utilization and health claim reimbursements, and 3) absenteeism and presenteeism.
Relative cost of different programs | ~1-3 years post baseline
  Determine the overall relative impact of STH+ and STH on net program costs.
Improvement in nutrition | ~1-2 years post baseline
  Determine whether employees participating in STH+ will experience greater improvements in diet, as measured by amount of calories consumed from fat and amount of fruits and vegetables consumed than employees in STH.

CONTACTS AND LOCATIONS:
Overall Officials: Truls Ostbye, MD, PHD, Principal Investigator — Duke University
Locations (1):
- Duke University Dept. of Community and Family Medicine, Durham, North Carolina, United States

REFERENCES:
- [Background] Ostbye T, Stroo M, Brouwer RJ, Peterson BL, Eisenstein EL, Fuemmeler BF, Joyner J, Gulley L, Dement JM. The steps to health employee weight management randomized control trial: rationale, design and baseline characteristics. Contemp Clin Trials. 2013 Jul;35(2):68-76. doi: 10.1016/j.cct.2013.04.007. Epub 2013 May 3. PMID 23648394
- [Result] Ostbye T, Stroo M, Brouwer RJ, Peterson BL, Eisenstein EL, Fuemmeler BF, Joyner J, Gulley L, Dement JM. Steps to Health employee weight management randomized control trial: short-term follow-up results. J Occup Environ Med. 2015 Feb;57(2):188-95. doi: 10.1097/JOM.0000000000000335. PMID 25654520
- [Result] Ostbye T, Stroo M, Eisenstein EL, Dement JM. The Effects of Two Workplace Weight Management Programs and Weight Loss on Health Care Utilization and Costs. J Occup Environ Med. 2016 Feb;58(2):162-9. doi: 10.1097/JOM.0000000000000586. PMID 26849260